CLINICAL TRIAL: NCT01095575
Title: Pre- vs. Post-Incisional Epidural Morphine: Higher Postoperative Pain Perception and Extra Morphine Consumption
Brief Title: Pre- Versus Post-Incisional Epidural Morphine: Higher Postoperative Pain Perception and Extra Morphine Consumption
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Weinbroum Avraham, Tel Aviv Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: weinbroum pain
Record Dates: First submitted 2010-03-28; First posted 2010-03-30 (Estimated); Last update posted 2010-04-12 (Estimated); Status verified 2010-03

CONDITIONS: Pain
Keywords: Epidural; Morphine; Preoperative; Postoperative; Analgesia; Tolerance; Preoperative, Postoperative Analgesia
MeSH Terms: conditions — Pain; Agnosia | interventions — Saline Solution; Morphine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- group 1 (Active Comparator): NS preoperatively and MO postoperatively
  Interventions: Drug: normal saline 3 ml, morphine 3mg
- group 2 (Active Comparator): MO preoperatively and NS postoperatively
  Interventions: Drug: normal saline 3 ml, morphine 3mg

INTERVENTIONS:
Drug: normal saline 3 ml, morphine 3mg — On the day of surgery, patients were brought to the operating room (OR) where routine monitors were placed and an epidural catheter was inserted at the level of L3-4 to a distance of 10 cm. All patients received two injections via the catheter: one injection contained 3 mg morphine (MO), and the other contained normal saline (NS) of the same volume. Patients were randomized to receive either NS preoperatively and MO postoperatively or vice versa. The first injection was administered 40 minutes before initiation of surgery, and the second one was given 15 minutes after surgery ended. All epidural catheters were removed before the patients were discharged from the post-anesthesia care unit (PACU).

SUMMARY:
Background and Objectives: Neuraxial administration of morphine is an effective way of controlling postoperative pain and reducing analgesic consumption. Several animal models have demonstrated that preemptive administration of neuraxial narcotics reduced pain while others revealed the induction of post-incisional hypersensitivity. There have been no consistent results in clinical setting either. This double blind, randomized study compared the effects of PRE- vs. POST-incisional administration of neuraxial morphine on postoperative pain perception and analgesic requirements over 48 hours following laparotomy for open colectomy under standardized general anesthesia.

Methods: Twenty patients received epidural morphine (3 mg) pre-incision and saline after wound closure (MO1 group), and 20 patients received epidural saline before incision and morphine after wound closure (MO2 group). Postoperatively, all patients received boluses of morphine (1.5 mg) via intravenous patient-controlled analgesia (IV-PCA), and rescue doses of intramuscular diclofenac (75 mg) every 6 hours, as needed.

ELIGIBILITY:
Inclusion Criteria:

1.adults scheduled for elective laparotomy and colon surgery with the duration of surgery expected to last for at least 2 hours.

Exclusion Criteria:

1. allergy to morphine, fentanyl, non-steroidal anti-inflammatory drugs or any of the intraoperative anesthetic medications
2. use of opioids, sedatives or stimulants during 21 days prior to surgery, psychiatric illness
3. congestive heart failure, respiratory failure, neuromuscular disease or presence of a chronic pain syndrome
4. Pregnant women and patients unable to sign their own consent form

Ages: 18 Years to 75 Years | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2006-01; Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Subjective pain intensity, using a visual analogue scale (VAS) from 0 (no pain) to 10 (unbearable pain) | 48 hours

SECONDARY OUTCOMES:
Consumption of analgesics | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Avraham Weinbroum, MD, Principal Investigator — Tel Aviv Medical Center